CLINICAL TRIAL: NCT06286137
Title: Duration of Music Interventions and PAiN Tolerance in Healthy Individuals: the DOMINANT Trial
Brief Title: Duration of Music Interventions and Pain Tolerance (DOMINANT)
Acronym: DOMINANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Markus Klimek, Vice-Chairman / Director Residency Training Program, Department of Anesthesiology, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL82922.078.22
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Pain, Acute
Keywords: Music-induced analgesia
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: The randomized controlled trial will have four study arms. Subjects will be assigned to one of the four arms: control without music and music groups with 1 minute, 5 minutes and 20 minutes. All subjects will receive electric stimuli in three phases. In each phase, subject will be exposed to three consecutive stimuli. First a detection threshold will be measured. Secondly a baseline test will be performed in order to assess basic levels of pain endurance. Hereafter, the intervention phase starts. Subjects in the music groups will listen to 1, 5 and 20 minutes of their own preferred music through headphones. Directly after, all subjects will again receive three electric stimuli.
Masking Description: Due to the nature of the study and the music intervention, it is not possible to blind participants and investigators. However, participants will not be informed of the study arm to which they are randomized in advance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (Active Comparator): The control group will be seated for 20 minutes without doing anything else, and not listen to music.
  Interventions: Other: Not listening to music
- 1 minute music group (Experimental): The 1 minute music group will be seated for 19 minutes without doing anything else, and listen to music for 1 minute.
  Interventions: Other: Listening to music for 1 minute
- 5 minutes music group (Experimental): The 5 minutes music group will be seated for 15 minutes without doing anything else, and listen to music for 5 minutes.
  Interventions: Other: Listening to music for 5 minutes
- 20 minutes music group (Experimental): The 20 minutes music group will listen to music for 20 minutes.
  Interventions: Other: Listening to music for 20 minutes

INTERVENTIONS:
Other: Listening to music for 1 minute — Participants will be instructed to make a 20-minute playlist with their own preferred music, using a tablet and a music listening app. That playlist will then be presented on shuffle mode for 1 minute through headphones provided by the hospital. Volume can be selected by the participants. However, in order to prevent hearing loss the volume cannot exceed 80 decibels. The 19 minutes before the 1 minute music listening intervention, participants will be instructed to remain seated and are not allowed to do anything else (for example using their phones).
  Arms: 1 minute music group
Other: Listening to music for 5 minutes — Participants will be instructed to make a 20-minute playlist with their own preferred music, using a tablet and a music listening app. That playlist will then be presented on shuffle mode for 1 minute through headphones provided by the hospital. Volume can be selected by the participants. However, in order to prevent hearing loss the volume cannot exceed 80 decibels. The 15 minutes before the 5 minutes music listening intervention, participants will be instructed to remain seated and are not allowed to do anything else (for example using their phones).
  Arms: 5 minutes music group
Other: Listening to music for 20 minutes — Participants will be instructed to make a 20-minute playlist with their own preferred music, using a tablet and a music listening app. That playlist will then be presented on shuffle mode for 20 minutes through headphones provided by the hospital. Volume can be selected by the participants. However, in order to prevent hearing loss the volume cannot exceed 80 decibels.
  Arms: 20 minutes music group
Other: Not listening to music — Participants will be instructed to remain seated and are not allowed to do anything else (for example using their phones), for a duration of 20 minutes.
  Arms: Control group

SUMMARY:
This study will investigate the effect of different durations of music interventions (1, 5 and 20 minutes of music) on pain tolerance.

DETAILED DESCRIPTION:
Music interventions reduce perioperative pain and anxiety. However, it is yet unclear how long music needs to be presented in order to have an effect. Therefore, the investigators would like to propose a pilot randomized controlled trial in order to investigate the optimal duration of musical interventions. The main objective of this study is to investigate the effect of different durations of music interventions on pain tolerance (expressed in amperage). Secondary objectives are to investigate the effects of music duration on heart rate variability (expressed in milliseconds) and subjective measurements of emotions, anxiety and pain. Healthy volunteers (age ≥18 years) will be included, and the study will take place at the outpatient clinic of the Center of Pain Medicine, Erasmus Medical Center, Rotterdam.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 64 years of age
* Sufficient knowledge of the Dutch language to understand the study documents (in the judgement of the attending physician or researcher)
* Provision of written informed consent by subject

Exclusion Criteria:

* Significant hearing impairment
* Current complaints of tinnitus
* Current use of analgesic medication
* Presence of acute or chronic pain
* History of cardiac disease or arrhythmias
* Current treatment by a medical specialist or general practitioner
* Professional musician or singer (practicing in average >1 hour each day)
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Pain tolerance | At the end of the intervention, after the 20 minutes of listening to music or sitting in silence. Measured at the same day as the experiment.
  The primary objective of the study is the pain tolerance. This tolerance will be measured using electric stimuli directly after the 20 minutes of listening to music or sitting in silence. Each measurement will be performed three times. Results will be expressed in amperage.

SECONDARY OUTCOMES:
Heart rate variability (HRV) | During the 20 minutes of listening to music or sitting in silence, and during the eletric stimuli directly after those 20 minutes. Measured at the same day as the experiment.
  HRV, the variation in time between adjacent heartbeats, can be used as a marker for autonomic function. Furthermore, an increase of HRV has been found after music interventions, possibly due to the effect on the parasympatic nervous system. HRV will be measured continuously using an Acentas Chest Strap (BM innovations GmbH).
Level of perceived anxiety, Spielberger State-Trait Anxiety Inventory (STAI)-6 questionnaire | At baseline and immediately after the intervention, after the electric stimuli. Measured at the same day as the experiment.
  The STAI-6 questionnaire is a validated and frequently used questionnaire to assess anxiety. The questionnaire comprises six items and the total scores ranges from 20 to 80, with a higher score indicating a higher level of anxiety.
Valence and arousal, Self-Assessment manikin (SAM) questionnaire | At baseline and immediately after the intervention, after the electric stimuli. Measured at the same day as the experiment.
  The SAM is a non-verbal pictorial assessment technique that directly measures the pleasure, arousal, and dominance associated with a person's affective reaction to a wide variety of stimuli. Each measurement value ranges from 1 to 9, which indicates different levels of pleasure, arousal and dominance.
Music listening Questionnaire | At baseline. Measured at the same day as the experiment.
  This questionnaire will consist of 7 open questions about music importance and music listening behavior. Participants will be asked to what extend they are a lover of music from a scale of 1 to 7, where a higher value is a higher amout of loving music. Next, participants will be asked how many minutes per day they listen actively and passively to music. Finally, participants will be asked in open questions about their favorite genres, their favorite moments of listening to music, if they play an instrument and if there is music that they dislike.
Pain intensity | At the end of the intervention, immediately after each electric stimulus. Measured at the same day as the experiment.
  Pain intensity will be measured using the Numeric Rating Scale. Values range from 0 to 10, with higher values indicating higher pain intensity.
Pain unpleasantness | At the end of the intervention, immediately after each electric stimulus. Measured at the same day as the experiment.
  Pain unpleasantness will be measured using the Numeric Rating Scale. Values range from 0 to 10, with higher values indicating higher pain unpleasantness.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Klimek, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will only be shared upon request. This decision will be made by the principal investigator.

REFERENCES:
- [Background] Kuhlmann AYR, de Rooij A, Kroese LF, van Dijk M, Hunink MGM, Jeekel J. Meta-analysis evaluating music interventions for anxiety and pain in surgery. Br J Surg. 2018 Jun;105(7):773-783. doi: 10.1002/bjs.10853. Epub 2018 Apr 17. PMID 29665028
- [Background] Fu VX, Oomens P, Klimek M, Verhofstad MHJ, Jeekel J. The Effect of Perioperative Music on Medication Requirement and Hospital Length of Stay: A Meta-analysis. Ann Surg. 2020 Dec;272(6):961-972. doi: 10.1097/SLA.0000000000003506. PMID 31356272
- [Background] Koelsch S. Brain correlates of music-evoked emotions. Nat Rev Neurosci. 2014 Mar;15(3):170-80. doi: 10.1038/nrn3666. PMID 24552785
- [Background] Basinski K, Zdun-Ryzewska A, Greenberg DM, Majkowicz M. Preferred musical attribute dimensions underlie individual differences in music-induced analgesia. Sci Rep. 2021 Apr 21;11(1):8622. doi: 10.1038/s41598-021-87943-z. PMID 33883585
- [Background] Valevicius D, Lepine Lopez A, Diushekeeva A, Lee AC, Roy M. Emotional responses to favorite and relaxing music predict music-induced hypoalgesia. Front Pain Res (Lausanne). 2023 Oct 25;4:1210572. doi: 10.3389/fpain.2023.1210572. eCollection 2023. PMID 38028433
- [Background] Howlin C, Stapleton A, Rooney B. Tune out pain: Agency and active engagement predict decreases in pain intensity after music listening. PLoS One. 2022 Aug 3;17(8):e0271329. doi: 10.1371/journal.pone.0271329. eCollection 2022. PMID 35921262
- [Background] Martin-Saavedra JS, Vergara-Mendez LD, Pradilla I, Velez-van-Meerbeke A, Talero-Gutierrez C. Standardizing music characteristics for the management of pain: A systematic review and meta-analysis of clinical trials. Complement Ther Med. 2018 Dec;41:81-89. doi: 10.1016/j.ctim.2018.07.008. Epub 2018 Jul 11. PMID 30477868
- [Background] Lunde SJ, Vuust P, Garza-Villarreal EA, Vase L. Music-induced analgesia: how does music relieve pain? Pain. 2019 May;160(5):989-993. doi: 10.1097/j.pain.0000000000001452. No abstract available. PMID 30507782